CLINICAL TRIAL: NCT05978570
Title: Assessing the Impact of Physical Therapy in the Pre-cystectomy Pathway in Patients With Bladder Cancer on Patient Outcomes
Brief Title: Physical Therapy in Pre-cystectomy Patients
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC2251
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Bladder Cancer
Keywords: radical cystectomy; physical therapy; exercise program
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A personally tailored exercise: A personally tailored exercise program will be offered to the participants after the Physical Therapy assessment, before the surgery.

SUMMARY:
This single-site, non-randomized, study evaluates the impact of a physical therapy consultation for patients with bladder cancer scheduled for radical cystectomy (RC). The purpose of this study is to investigate whether consultation with a physical therapist and the development of a personally tailored exercise program in the pre-cystectomy period for patients with bladder cancer will result in reduced post-operative complications, morbidity, length of inpatient stay, improve readmission 30-day and 90-day and improve 90-day mortality. This study will be partially retrospective (pre-implementation of a physical therapy consultation order) and partially prospective.

ELIGIBILITY:
In order to participate in this study a subject must meet all of the eligibility criteria outlined below:

Inclusion Criteria:

1. Age ≥ 18 years at the time of bladder cancer diagnosis
2. History of bladder cancer
3. Performance of radical cystectomy

Exclusion Criteria:

1. No history of bladder cancer or radical cystectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are with bladder cancer and receiving treatment at the study site.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2023-08-27 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Thirty-day readmission rates | Up to 30 days after the date of cystectomy
  Thirty-day readmission rates will be defined as the comparison of the number of hospital admission after physical therapy consultation and tailored exercises and historical hospital admission data.

SECONDARY OUTCOMES:
The proportion of individuals who received a physical therapy consultation | 1 day (the date of cystectomy)
  The feasibility of implementing a physical therapy consultation and tailored exercise program in the pre-cystectomy treatment pathway will be determined by calculating the proportion of individuals who received a physical therapy consultation in the prospective group.
Ninety-day readmission rates | Up to 90 days after the date of cystectomy
  Ninety-day readmission rates will be defined as the comparison of the number of hospital admission after physical therapy consultation and tailored exercises and historical hospital admission data.
Acute care length of stay | Starting to the exercises to up to 90 days after the date of cystectomy
  Acute care length of stay will be defined as comparing number of hospital day stay after physical therapy consultation and tailored exercises and historical hospital admission data.
Mortality rates | Up to 90 days after the date of cystectomy
  Mortality rates will be defined as the comparison of the number of subjects who died after physical therapy consultation and tailored exercises and historical hospital admission data.
Post-cystectomy complication types and rates | Up to 90 days after the date of cystectomy
  Post-cystectomy complication types and rates will be defined as comparison of the numbers and types of complications after physical therapy consultation with tailored exercises and historical data.

CONTACTS AND LOCATIONS:
Overall Officials: Sasha Knowlton, Principal Investigator — Lineberger Comprehensive Cancer Center, The University of North Carolina Chapel Hill
Locations (1):
- Lineberger Comphrehensive Cancer Center at University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials